CLINICAL TRIAL: NCT01675570
Title: A Phase II, Multi-Center, Randomized, Placebo-Controlled, Double-Masked Study of RX-10045 (0.09%) in the Treatment of Dry Eye Disease
Brief Title: A Study of RX-10045 in the Treatment of Dry Eye Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: C.T. Development America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CTD1201
Record Dates: First submitted 2012-08-28; First posted 2012-08-30 (Estimated); Last update posted 2013-02-08 (Estimated); Status verified 2013-02

CONDITIONS: Dry Eye Syndrome
Keywords: RX-10045; Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes | interventions — isopropyl 5,12-hydroxypentadeca-8,10-dien-6,14-diynoate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RX-10045 active arm (Experimental): RX-10045 Opththalmic Solution, 0.09%
  Interventions: Drug: RX-10045
- Vehicle for RX-10045 arm (Placebo Comparator): Vehicle of RX-10045 Ophthalmic Solution
  Interventions: Drug: Vehicle for RX-10045

INTERVENTIONS:
Drug: RX-10045 — One drop of RX-10045 ophthalmic solution will be instilled in each eye, twice a day, approximately 12 hours apart for 28 days.
  Arms: RX-10045 active arm
Drug: Vehicle for RX-10045 — One drop of RX-10045 placebo solution will be instilled in each eye, twice a day, approximately 12 hours apart for 28 days.
  Arms: Vehicle for RX-10045 arm

SUMMARY:
The primary purpose of this study is to assess the efficacy, tolerability and safety of RX-10045 Ophthalmic Solution in patients with Dry Eye Disease.

ELIGIBILITY:
Inclusion Criteria:

1. Have a patient reported history of dry eye in both eyes
2. Presence of dry eye symptoms
3. Presence of dry eye signs, destabilized tear film break-up time and corneal staining

Exclusion Criteria:

1. Known contraindications or sensitivities to study medication or its components
2. Any ocular condition that, in the opinion of the investigator, could affect the subject's safety or trial parameters
3. Use of disallowed medication during the period indicated prior to the enrollment or during the study
4. Be a female who is currently pregnant, planning a pregnancy, lactating, or not using a medically acceptable form of birth control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2012-08; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Corneal staining | Baseline to day 28
Worst symptom score | Baseline to day 28

SECONDARY OUTCOMES:
Ocular discomfort symptom score | Baseline to day 28
Tear film break-up time | Baseline to day 28
Visual-related function subscale of Ocular Surface Disease Index score | Baseline to day 28

CONTACTS AND LOCATIONS:
Overall Officials: Gail Torkildsen, MD, Principal Investigator — Andover Eye Associates
Locations (1):
- Andover Eye Associates, Andover, Massachusetts, United States